CLINICAL TRIAL: NCT07391111
Title: THE EFFECT OF STANDARD PATIENT AND WEB-BASED SIMULATION APPLICATIONS ON NURSING STUDENTS' KNOWLEDGE AND ATTITUDES TOWARDS FALLS
Brief Title: THE EFFECT OF STANDARD PATIENT AND WEB-BASED SIMULATION ON FALL KNOWLEDGE AND ATTITUDES AMONG NURSING STUDENTS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ESRA ERTUĞRUL (Other)
Responsible Party: Sponsor-Investigator, ESRA ERTUĞRUL, Lecturer, Aydin Adnan Menderes University
Organization: Aydin Adnan Menderes University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2024/028
Record Dates: First submitted 2025-12-31; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Patient Safety; Fall; Simulation Edication
Keywords: web-based simulation; standard patient; nursing students; randomized controlled trial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 Group trained with a standard patient in the simulation lab (Experimental)
  Interventions: Other: Standardized patient
- Group 2 The group is receiving web-based simulation training in a laboratory setting. (Experimental)
  Interventions: Other: web-based simulation
- Group 3 Classical classroom education group. (No Intervention)

INTERVENTIONS:
Other: Standardized patient — The group receiving training with standard patients in a simulation laboratory environment.
  Arms: Group 1 Group trained with a standard patient in the simulation lab
Other: web-based simulation — Group receiving training through web-based simulation in a laboratory environment.
  Arms: Group 2 The group is receiving web-based simulation training in a laboratory setting.

SUMMARY:
The most fundamental principle of any healthcare service is "First, do no harm." No one should be harmed in healthcare services. Falls are the most frequently reported and preventable incident among all safety incidents in the hospital environment. However, falls are the most frequently reported incident among all safety incidents. Patient falls are the most common adverse events in hospitals. Patient falls in hospitals cause physiological and psychological harm to patients, affect the timeliness, effectiveness, and efficiency of care, and lead to increases in hospital costs and length of stay. Therefore, preventing falls, which have serious consequences, is of vital importance in terms of patient safety and healthcare quality. Nurses are a group that can sensitively identify and manage issues related to patient safety. Therefore, it is important to identify and reduce the underlying risk factors for falls in patients and to provide appropriate nursing interventions to prevent secondary injuries in patients who have fallen.

Simulation is an important part of nursing education because it improves patient care and ensures patient safety. Simulation-based learning provides students with realistic clinical situations, allowing them to practice clinical skills in a safe environment. This enables students to develop their clinical skills, communication, decision-making, and self-efficacy in a risk-free, safe, and structured environment, representing a contemporary teaching approach.

Teaching safe patient care during nursing students' education is one of the most fundamental elements of nursing education. Inadequate nursing knowledge and attitudes increase the risk of falls among patients receiving care. Students with insufficient clinical experience are at high risk of making undesirable errors in patient care. It is important to increase nursing students' knowledge and attitudes regarding falls during their education.

The standard patient and web-based simulation application offers the closest experience to real clinical situations, providing students with significant potential to become aware of falls they may encounter in practice and prevent potential errors. The increasing importance given to patient safety due to the rising number of fall cases supports the necessity of this research. The aim of this study is to evaluate the effect of standard patient and web-based simulation methods on nursing students' knowledge and attitudes regarding falls.

ELIGIBILITY:
Inclusion Criteria:Students were included in the study if they were:

* A senior nursing student at Aydın Adnan Menderes University Faculty of Nursing
* Volunteering to participate in the study
* Not absent at any time during the study period
* Working/not working as a nurse

Exclusion Criteria:

* Graduated from a health vocational high school
* Admitted through the Foreign Student Exam (YÖS)
* Graduated from a health-related associate's degree program and then enrolled in the nursing department through the Vertical Transfer Exam (DGS)
* Students who did not wish to participate in the study were excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-22 (Estimated)

PRIMARY OUTCOMES:
Planned Mean Change in Total Knowledge Score on the Fall Prevention Knowledge Test (0-28) | From enrollment to the 8th week of the intervention
  Planned Mean Change in Total Knowledge Score on the Fall Prevention Knowledge Test (0-28) Total knowledge score will be measured using the Fall Prevention Knowledge Test among nursing students. Change from baseline will be assessed.
Planned Mean Change in Attitude Score on the Nurses' Attitudes Toward Fall Prevention Scale | From enrollment to 8 weeks after intervention
  Planned Mean Change in Attitude Score on the Nurses' Attitudes Toward Fall Prevention Scale Mean attitude score will be measured using the Nurses' Attitudes Toward Fall Prevention Scale among nursing students. Change from baseline will be assessed.

SECONDARY OUTCOMES:
Planned Mean Change in Total Knowledge Score on the Patient Fall Prevention Knowledge Test | Immediately after the intervention
  The change in the total knowledge scores of nursing students will be measured using the Patient Fall Prevention Knowledge Test. Change from baseline will be assessed.
Planned Mean Change in Average Attitude Score on the Nurses' Attitudes Towards Fall Prevention Scale | Immediately after the intervention
  The change in the average attitude scores of nursing students will be measured using the Nurses' Attitudes Towards Fall Prevention Scale. Change from baseline will be assessed.
Planned Mean Change in Student Satisfaction Score Regarding the Simulation Experience | Immediately after the intervention
  The change in the average satisfaction score of nursing students in the experimental group will be measured using the Student Satisfaction Scale. Change from baseline will be assessed.
Planned Mean Change in Learning Self-Confidence Score Regarding the Simulation Experience | Immediately after the intervention
  The average learning self-confidence score of nursing students in the experimental group will be measured using the Learning Confidence Scale. Change from baseline will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Adnan Menderes University, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
This study does not plan to share raw data at the individual level. However, to promote transparency of research findings, summary data (demographic characteristics, pretest and posttest scores, group comparisons, and analysis results) that do not include participant identification will be shared with researchers upon request. No personal identifying information (name, contact information, institutional information, etc.) will be shared.
Supporting Information: SAP, ICF, CSR
Time Frame: August 2026-December 2026
Access Criteria: Access to data will be available only after a written request from the researcher and a review by the research team for scientific relevance. Access will only be provided by securely transmitting designated datasets via email; no sharing will be made via any open-access repository or online platform.